CLINICAL TRIAL: NCT03815448
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial of Methotrexate (MTX) in the Treatment of Advanced Knee Osteoarthritis With Effusion-synovitis
Brief Title: Methotrexate in the Treatment of Advanced Knee Osteoarthritis With Effusion-synovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Beijing Hospital (Other Government); Xuanwu Hospital, Beijing (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Second People's Hospital of GuangDong Province (Other); Peking University People's Hospital (Other); Shenzhen Third People's Hospital (Other); Central People's Hospital of Zhanjiang (Other); Qingyuan People's Hospital (Other)
Responsible Party: Principal Investigator, Ding Changhai, Director,Clinical Research Center, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-FSMYK-001
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis; Effusion Synovial; Knee Pain
Keywords: Methotrexate; knee osteoarthritis; Magnetic Resonance imaging; pain; synovitis
MeSH Terms: conditions — Osteoarthritis, Knee; Hydrarthrosis; Pain; Synovitis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Experimental): Methotrexate 2.5mg/ tablet, oral, once a week, 2-6 tablets each time
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Placebo 2.5mg/ tablet,oral,once a week,2-6 tablets each time
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methotrexate — Participants randomized to methotrexate group will receive active drug, methotrexate. Starting from 5 mg/week, the dosage will be adjusted to 10 mg/week if the participants can tolerate for 2 weeks. After 2 weeks, the dosage will be adjusted to 15 mg/week until the end of the study if the participants can tolerate.
  Other Names: MTX
  Arms: Methotrexate
Other: Placebo — Participants randomized to placebo group will receive placebo tablets. Starting from 5 mg/week for 2 weeks, the dosage will be adjusted to 10 mg/week; after 2 weeks, the dosage will be adjusted to 15 mg/week until the end of the study.
  Arms: Placebo

SUMMARY:
This multicentre randomized placebo-controlled clinical trial aims to evaluate whether methotrexate (MTX) has effects of relieving symptoms and reducing inflammation on advanced knee osteoarthritis (OA) with inflammatory phenotype. Participants will be randomly allocated to either MTX group or placebo group receiving MTX or placebo once a week. The primary outcomes are effusion-synovitis volume measured by magnetic resonance imaging (MRI) and knee pain assessed by visual analogue scale (VAS).

DETAILED DESCRIPTION:
OA is a common chronic musculoskeletal disease in middle-aged and elderly people, which is characterized by loss of articular cartilage and other structural damage of joints. Currently, there is no effective treatment to reduce disease severity and progression of knee OA, particularly in mid to late-stages. Analgesics and anti-inflammatory drugs can only have effects in a short time, with obvious side effects, and are not effective for all patients. In the late stage, most patients are performed with arthroplasty. However, arthroplasty is expensive and has high technical requirements for surgeons. Therefore, it is urgent to find effective drugs or means to control the symptoms and disease progression of knee OA.

Due to different etiologies, OA may have different clinical phenotypes, one of which is mainly manifested by synovitis and is common in patients with advanced OA. Pathological studies have shown that OA synovitis is significantly related to adjacent cartilage lesions, and its pathological changes were similar to rheumatoid arthritis (RA), but the degree of the latter is relatively mild. MTX can alleviate joint inflammation and delay joint structural damage. In patients with rheumatoid arthritis, MTX can reduce suprapatellar bursa synovitis by 35%, inhibit the inflammatory response of synovial tissue, including reducing the number of macrophage, inhibiting the expression of intercellular adhesion molecule -1, interleukin (IL)-1, tumour necrosis factor (TNF)-α and C-reactive protein (CRP), and even reduce bone marrow lesions (BMLs) and synovitis in very early stages. In patients with early-stage undifferentiated arthritis, MTX treatment for two months can significantly reduce synovitis and exudation, alleviate BMLs and reduce serum CRP level. Chronic calcium pyrophosphate deposition disease is a non-autoimmunity inflammatory arthritis which can be followed by more severe OA. After 6-81 months of treatment with MTX (5-20 mg/week), the pain intensity, swelling and the number of involved joints were significantly decreased. Based on all the evidence as discussed above, MTX may have beneficial effects on OA via a variety of mechanisms, including reduction of synovitis and effusion, and decreases in inflammatory cytokines.

The investigators design a multicentre randomized placebo-controlled clinical trial over 12 months. The aim is to determine if MTX can relieve symptom and reduce effusion-synovitis in patients with advanced knee OA. The investigators will recruit 200 participants who are in the advanced stage of symptomatic knee OA with effusion-synovitis grade of ≥ 2 (assessed by MRI). Participants will be randomly allocated to MTX group (start from 5 mg per week for the first two weeks and increase to 10 mg per week for the second two weeks and 15 mg per week for the remaining period if tolerated) or placebo group. Intention to treat and per protocol analyses of primary and secondary outcomes will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Meet the America College of Rheumatology (ACR) criteria for clinical knee OA assessed by a rheumatologist
* Knee pain, visual analogue scale (VAS) pain at least 40mm
* Kellgren-Lawrence(K-L) grade of 2-4
* Physical examination showed signs of inflammation (at least 2 of the following 4 clinical signs of inflammation: warmth around the joint; tenderness around joint margin; articular cavity effusion; swelling of soft tissue around the knee joint)
* MRI evaluated effusion synovitis grade of ≥ 2
* Capable of understanding the study requirements and willing to cooperate with study instructions, and voluntarily sign informed consent

Exclusion Criteria:

* Inflammatory arthritis (such as gout, reactive arthritis, rheumatoid arthritis, psoriatic arthritis, seronegative spondyloarthropathy), systemic lupus erythematosus
* Knee surgery or arthroscopic examinations were performed or planned within one year, Severe valgus knee deformity (angle of genu valgum > 30°) or previous traumatic history
* MRI contraindications
* Intra-articular injection, intramuscular injection or oral glucocorticoid were used within the last 4 weeks
* Other anti-synovitis agents (such as hydroxychloroquine and sulfasalazine) were applied in the past 3 months
* Clinical significant conditions, such as (but not limited to) active malignant tumor, abnormal renal function (assessed by GFR), hepatic abnormalities [active hepatitis B, hepatitis C, abnormal liver function (ALT is more than twice the upper limit)], respiratory diseases (lung infection, pulmonary fibrosis), hematological changes (e.g white blood cell (WBC) count < 4 x 10^9 /L, platelet < 100 x 10^9 /L or hemoglobin < 100 g/L), serious diseases of gastrointestinal, endocrine, heart, nerve or brain assessed by clinical physicians
* Infectious history such as HIV infection
* Hypersensitivity to methotrexate
* Pregnant and Lactating women

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Effusion-synovitis | 12 months
  Knee effusion-synovitis volume/maximal area at suprapatellar pouch will be measured, and severity will be scored from 0-3 in terms of the estimated maximal distension of the synovial cavity by assessing the amount of intra-articular fluid-equivalent signal on T2-weighted MRI. Effusion at central portion, posterior femoral recess and subpopliteal recess will also be assessed.
VAS knee pain | 12 months
  Knee pain will be assessed by a 100mm VAS with terminal descriptors of "no pain" and "worst pain possible".

SECONDARY OUTCOMES:
Infrapatellar fat pad (IPFP) signal intensity alteration | 12 months
  Signal intensity alterations with IPFP was defined as discrete areas of increased signal. Standard deviation of IPFP signal intensity and Clustering Factor was used to represent the signal intensity alteration with IPFP.
Western Ontario and McMaster Universities Index (WOMAC) total score | 12 months
  WOMAC is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain (5 items), stiffness (2 items) and physical function (17 items).The score is higher, the knee function is worse.
Outcome Measures in Rheumatology Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) responders | 12 months
  The OMERACT-OARSI consists outcome measures in rheumatology arthritis clinical trials including pain, functional impairment and patient's global assessment. For each of these domains, a response was defined by both relative and an absolute change.

CONTACTS AND LOCATIONS:
Overall Officials: Changhai Ding, MD, Principal Investigator — Clinical Research Center of Zhujiang Hospital
Locations (11):
- China (11):
  - The 1st Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Hospital, Beijing, Guangdong
  - Zhujiang Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Second People's Hospital of Guangdong Province, Guanzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - The Third Hospital of Shenzhen, Shenzhen, Guangdong
  - Central People's Hospital of Zhanjiang, Zhanjiang, Guangdong
  - Peking University People's Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking Union Medical College University, Beijing

REFERENCES:
- [Derived] Zhu Z, Yu Q, Leng X, Xu J, Ren L, Wang K, Huang C, Pan Y, Zhao Y, Li T, Mei Y, Guan M, Li X, Zhang Z, Wu J, Chen Y, Qu Y, Zhu X, Liao Q, Wang Z, Liao Z, Xi Y, Deng W, Wang K, Zhu T, Zhang Y, Gao L, Zhou X, Han W, Ruan G, Zhang Y, Cao P, Gao P, Chen H, Dang Q, Cicuttini FM, Hunter DJ, Li Z, Zeng X, Ding C. Low-Dose Methotrexate for the Treatment of Inflammatory Knee Osteoarthritis: A Randomized Clinical Trial. JAMA Intern Med. 2025 Jul 1;185(7):808-816. doi: 10.1001/jamainternmed.2025.1359. PMID 40455462
- [Derived] Liu Q, Ren J, Zhang W, Liang T, Wang Z, Xie S, Li Y, Hou J, Wang K, He R. Measured Resection as Gap Balance Method in Mobile-Bearing Medial Unicompartmental Knee Arthroplasty: A Randomized Controlled Trial. Orthop Surg. 2025 Feb;17(2):603-613. doi: 10.1111/os.14346. Epub 2025 Jan 5. PMID 39757775
- [Derived] Zhu Z, Yu Q, Leng X, Han W, Li Z, Huang C, Gu J, Zhao Y, Wang K, Li T, Mei Y, Xu J, Zhang Z, Hunter D, Cicuttini F, Zeng X, Ding C. Can low-dose methotrexate reduce effusion-synovitis and symptoms in patients with mid- to late-stage knee osteoarthritis? Study protocol for a randomised, double-blind, and placebo-controlled trial. Trials. 2020 Sep 16;21(1):795. doi: 10.1186/s13063-020-04687-3. PMID 32938470